CLINICAL TRIAL: NCT00232895
Title: Pain of Injection of Lipuro Propofol in Children Aged 1-7 Years
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Child Health (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 02AR36
Record Dates: First submitted 2005-10-04; First posted 2005-10-05 (Estimated); Last update posted 2007-03-28 (Estimated); Status verified 2007-03

CONDITIONS: ASA 1-2 Requiring Intravenous Cannulation for General Anaesthesia
MeSH Terms: interventions — Propofol

INTERVENTIONS:
Drug: lipuro propofol
Drug: standard formulation propofol

SUMMARY:
Randomised controlled trial of pain of injection of lipuro in children age 1-7 versus the pain of injection of the standard formulation

ELIGIBILITY:
Inclusion Criteria:

* ASA 1 or 2 requiring intravenous general anaesthetic

Exclusion Criteria:

-

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Study Completion 2005-08

PRIMARY OUTCOMES:
pain scores on induction of anaesthesia with propofol

CONTACTS AND LOCATIONS:
Overall Officials: Mark Thomas, Dr, Principal Investigator — Great Ormond Street Hospital
Locations (1):
- Great Ormond Street Hospital, London, United Kingdom